CLINICAL TRIAL: NCT07123233
Title: Reprocessing The Fear Of Pain - A Cognitive-Behavioral Protocol For Chronic Primary Orofacial Pain Diseases.
Brief Title: An Innovative Cognitive-Behavioral Treatment For Chronic Orofacial Pain
Acronym: FACE-PRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FACE-PRT; GR2024 (Other Grant/Funding Number: FONDAZIONE CARIPLO)
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Primary Orofacial Pain (CPOP); Persistent Idiopathic Facial Pain (PIFP)
Keywords: Cognitive-behavioral therapy; Pain-Reprocessing Therapy; Chronic Primary Orofacial pain; chronic pain; chronic primary pain; nociplastic pain
MeSH Terms: conditions — Chronic Pain; Nociplastic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRT-TAU (Experimental): Patients will attend 8 sessions of PRT treatments while undergoing their usual pharmacological treatment
  Interventions: Behavioral: Pain Reprocessing Therapy
- TAU (Placebo Comparator): Patients will undergo the usual pharmacological treatment.
  Interventions: Behavioral: Usual Therapy

INTERVENTIONS:
Behavioral: Pain Reprocessing Therapy — One cohort of 30 patients (PRT+TAU group) will receive eight sessions of Pain Reprocessing Therapy (PRT) in addition to Treatment-as-Usual (TAU). PRT is a cognitive-behavioral-inspired approach aimed at helping patients reinterpret chronic pain as brain-generated rather than structurally caused.
  A second cohort of 30 patients (TAU group) will undergo the same assessment phases but will receive only Treatment-as-Usual without PRT.
  Use this module to add a description of each group or cohort in the study and to list any interventions of interest.
  Arms: PRT-TAU
Behavioral: Usual Therapy — Patients undergo yhe usual pharmacological tretment as prescrived by neurologist
  Arms: TAU

SUMMARY:
Use these resources to provide understandable information about this study to patients, families, and health care providers:

The present randomized clinical trial (RCT), conducted at the IRCCS Carlo Besta Neurological Institute, aims to evaluate the effectiveness of Pain Reprocessing Therapy (PRT), a form of psychological support/psychotherapy based on cognitive-behavioral therapy, which has already proven effective in the treatment of other types of primary chronic pain.

Chronic Primary Orofacial Pain (CPOP) is a rare and complex form of chronic pain that predominantly affects adult women and occurs without evident lesions, yet has a significant emotional and functional impact. It was recently classified among chronic primary pain conditions in the ICD-11 and is considered a form of nociplastic pain, associated with alterations in brain connectivity. At present, pharmacological treatments have shown limited effectiveness.

This randomized clinical trial (RCT), conducted at the IRCCS Carlo Besta Neurological Institute, aims to evaluate the effectiveness of Pain Reprocessing Therapy (PRT), a form of psychological support/psychotherapy based on cognitive-behavioral therapy, which has already proven effective in the treatment of other types of primary chronic pain.

Sixty participants, all diagnosed with CPOP according to ICD-11 criteria, will be selected and randomly assigned to two groups: one will receive PRT, the other will receive treatment as usual (TAU).

The primary outcome of the study is the assessment of pain intensity reduction. Secondary outcomes include a broad range of psychosocial variables: improvement in quality of life, reduction of anxiety-depressive symptoms, catastrophizing, and other psychopathological traits. The effects of the therapy on brain connectivity will also be analyzed using fMRI, and on pain neurophysiology through the Conditioned Pain Modulation (CPM) paradigm. The protocol provides for the evaluation of therapy effectiveness at three follow-ups (3, 6, and 12 months) in order to measure the duration of effects.

Finally, through advanced statistical analysis tools and the support of artificial intelligence, the study also aims to identify specific clinical-neurofunctional profiles that may be useful for differential diagnosis and for tailoring therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Primary Orofacial Pain (CPOP) according to ICD-11 criteria.
* Patient-reported pain rating of 4 or higher out of 10 on the Brief Pain Inventory (BPI) question assessing average pain over the past week, consistent with inclusion criteria from previous chronic pain studies.
* Written informed consent.
* Age 18 years or older.

Exclusion Criteria:

* Age over 70 years.
* Current use of immunosuppressive medications (e.g., steroids).
* History of cancer (breast, thyroid, prostate, blood cancers, etc.).
* History of stroke, neurosurgical interventions, or brain tumors.
* History of specific inflammatory diseases (lupus, scleroderma, rheumatoid arthritis, polymyalgia rheumatica).
* History of psychiatric disorders such as schizophrenia, personality disorders, dissociative identity disorder, or other severe psychoses.
* Unexpected or unintentional weight loss of 10 kg or more in the year prior to recruitment.
* Difficulty participating due to logistical problems.
* Contraindications to undergoing functional magnetic resonance imaging (fMRI).
* Psychotherapy treatment of any kind within 15 months prior to the assessment date.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Average pain intensity over the past week. | 12 months
  Average pain intensity over the past week, measured using the Brief Pain Inventory-Short Form (BPI-SF). Score range: 0-10, with higher scores indicating greater pain intensity (worse outcome).

SECONDARY OUTCOMES:
Quality of life (EUROHIS-8) | 12 months
  It includes 8 items scored from 1 to 5 using a 5-point Likert scale investigating the satisfaction on different life domains (i.e., socio-economic conditions, health conditions, satisfaction with oneself and with one's relationships, etc.). A high total score corresponds to a high perception of quality of life.
Depressive and anxiety symptoms (BDI-II, BAI) | 12 months
  BDI-II - It consists of 21 items, each scored on a 4-point Likert scale (ranging from 0 to 3). A score above 13 points indicates the presence of clinical depression symptoms. BAI - It consists of 21 items, each scored on a 4-point Likert scale (ranging from 0 to 3). A score above 7 points indicates the presence of clinical anxiety symptoms.
Catastrophism (PCS) | 12 months
  it measures feelings of helplessness, magnification, and rumination. It has 13 items, each reflecting different aspects of catastrophic thinking related to pain. Respondents rate each item on a 5-point Likert scale, ranging from 0 (not at all) to 4 (extremely), based on how frequently they experience the thought or feeling described. Higher scores indicate greater levels of pain catastrophizing.
Psychopathology (MCMI-III) | 12 months
  It is a validated self-administered inventory with 175 true-false questions, assessing 14 personality disorder scales, divided into fourteen clinical patterns of personality based on Axis II disorders of DSM-IV, and ten clinical syndrome scales based on Axis I disorders of DSM-IV.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Grazzi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt S, Muhlan H, Power M. The EUROHIS-QOL 8-item index: psychometric results of a cross-cultural field study. Eur J Public Health. 2006 Aug;16(4):420-8. doi: 10.1093/eurpub/cki155. Epub 2005 Sep 1. PMID 16141303
- [Background] Monticone M, Baiardi P, Ferrari S, Foti C, Mugnai R, Pillastrini P, Rocca B, Vanti C. Development of the Italian version of the Pain Catastrophising Scale (PCS-I): cross-cultural adaptation, factor analysis, reliability, validity and sensitivity to change. Qual Life Res. 2012 Aug;21(6):1045-50. doi: 10.1007/s11136-011-0007-4. Epub 2011 Sep 13. PMID 21912846
- [Background] Benoliel R, Svensson P, Evers S, Wang SJ, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic secondary headache or orofacial pain. Pain. 2019 Jan;160(1):60-68. doi: 10.1097/j.pain.0000000000001435. PMID 30586072
- [Background] Robson WL, Leung AK, Kabani AM, Fick GH. Pseudohyperkalaemia in Kawasaki disease. Eur J Pediatr. 1993 Apr;152(4):379-80. doi: 10.1007/BF01956763. No abstract available. PMID 8482298
- [Background] Benoliel R, Gaul C. Persistent idiopathic facial pain. Cephalalgia. 2017 Jun;37(7):680-691. doi: 10.1177/0333102417706349. Epub 2017 Apr 20. PMID 28425324
- [Background] Nicholas M, Vlaeyen JWS, Rief W, Barke A, Aziz Q, Benoliel R, Cohen M, Evers S, Giamberardino MA, Goebel A, Korwisi B, Perrot S, Svensson P, Wang SJ, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic primary pain. Pain. 2019 Jan;160(1):28-37. doi: 10.1097/j.pain.0000000000001390. PMID 30586068